CLINICAL TRIAL: NCT00368836
Title: Expired CO2/O2 Analysis to Diagnose Pulmonary Embolism
Brief Title: Breath Analysis Technique to Diagnose Pulmonary Embolism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); WFD Ventures Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 433; R42HL086316-01 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2021-06-30 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Embolism
Keywords: Capnography; Thromboembolism; Arthroplasty; D-dimer
MeSH Terms: conditions — Pulmonary Embolism; Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BreathScreen PE + D-dimer (Experimental): CO2/O2 ratio will be measured using the Breath Screen PE device. D-dimer levels will also be collected.
  Interventions: Device: BreathScreen PE

INTERVENTIONS:
Device: BreathScreen PE — One minute of breath collection by tidal breathing into the BreathScreen PE and blood draw for D-dimer level

SUMMARY:
A pulmonary embolism (PE) is a blockage in one of the arteries of the lungs, and is usually caused by a traveling blood clot. The D-dimer blood test is currently used to diagnose PEs, but it is not always accurate for individuals who have recently undergone surgery or who have inflammatory-provoking diseases. The purpose of this study is to evaluate the effectiveness of the Carboximeter, a new PE diagnostic device that measures carbon dioxide (CO2) and oxygen (O2) output, in individuals at risk for developing PEs.

DETAILED DESCRIPTION:
PE is the second leading cause of sudden, unexpected death in the United States. In 90% of the cases, it is caused by deep vein thrombosis: a blood clot forms in a vein, travels through the bloodstream, and lodges in the lungs. PE symptoms vary, and can include cough, shortness of breath, chest pain, rapid breathing, or increased heart rate. Some medical procedures and diseases activate inflammation and blood coagulation, thereby making individuals more vulnerable to PE. Surgery, kidney dialysis, cancer, connective tissue diseases, infectious diseases, and being over 70 years old put individuals at increased risk for developing PEs. A common screening test for PE is the D-dimer blood test, which measures the level of a specific protein that is released following a PE. This test, however, has proven to be an unreliable diagnostic tool for individuals who are at high risk for PE. A more reliable diagnostic tool is needed. The Carboximeter is a new device that measures the ratio of CO2/O2 pressure in an individual's expired breath. By monitoring these components, researchers may be able to accurately diagnose PEs in high risk individuals. The purpose of this study is to evaluate the effectiveness of the Carboximeter at diagnosing PE in individuals at risk for developing PEs.

This study will be conducted in two phases. In Phase I, CO2/O2 ratio and D-dimer levels will be measured prior to and following orthopedic or cancer-related surgery in 100 individuals at risk for developing PEs. In Phase II, the same measurements will be carried out on 350 high risk individuals who are experiencing PE symptoms. These individuals will also undergo computed tomography (CT) angiography and venography, in which blood flow will be visualized using x-rays. A follow-up evaluation will occur 30 days later. If any participant from Phase I or II experiences a PE or a medical condition that affects their lungs, such as asthma or chronic obstructive pulmonary disease (COPD), researchers may schedule a follow-up evaluation to obtain repeat measurements.

ELIGIBILITY:
Phase I Inclusion Criteria:

* Experienced or is scheduled for at least one of the following:

  1. Hip or knee replacement surgery
  2. Hip or acetabular fracture surgery
  3. Pelvic fracture
  4. Decompression for spinal stenosis surgery
  5. Scoliosis corrective surgery
  6. Craniotomy surgery for brain tumor
  7. Surgery for any of the following cancers: bladder, colon (including caecum and rectum), kidney, ovary, pancreas, or uterus

Phase I Exclusion Criteria:

* Currently undergoing treatment for PE or has received treatment for PE in the 4 weeks prior to study entry
* Hospitalized for fewer than 2 days
* Anatomic abnormality that would prevent use of a mouthpiece
* Living situation that makes follow-up difficult (e.g., homeless, incarcerated)

Phase II Inclusion Criteria:

* Clinical suspicion of PE with signs or symptom suggestive of PE within 24 hours of presentation and at least one risk factor for PE, as defined under the criteria as outlined in this protocol
* CTA of pulmonary arteries ordered by clinical care providers
* 18 years or older or an emancipated 17 year old
* Written informed consent

Phase II Exclusion Criteria:

* Hemodynamic instability, including patients with a systolic blood pressure less than 90 mm Hg
* Severe respiratory distress or the inability to breathe room air without the sensation of severe dyspnea
* Pulse oximetry reading that declines more than 10% when exogenous oxygen is discontinued with accompanying worsening or new dyspnea
* Intubated
* Cannot breathe through the mouth owing to anatomic, physical or mental limitation
* No fixed address, no telephone number, are from out of town or have other reason to suspect difficulty with follow-up
* Incarceration
* Known active tuberculosis
* Prior PE or DVT with history of medical noncompliance with oral anticoagulation therapy based upon a history of unplanned subtherapeutic INR measurements (less than 1.5)
* Active PE within previous 6 months and currently under treatment with anticoagulation
* Pregnant
* Disallowed medications: treatment with any fibrinolytic agent within 48 hours prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jefferey A. Kline, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Kline JA, Hogg M. Measurement of expired carbon dioxide, oxygen and volume in conjunction with pretest probability estimation as a method to diagnose and exclude pulmonary venous thromboembolism. Clin Physiol Funct Imaging. 2006 Jul;26(4):212-9. doi: 10.1111/j.1475-097X.2006.00672.x. PMID 16836693
- [Derived] Kline JA, Watts J, Courtney D, Lee YY, Hwang S. Severe pulmonary embolism decreases plasma L-arginine. Eur Respir J. 2014 Mar;43(3):906-9. doi: 10.1183/09031936.00171913. Epub 2013 Nov 14. No abstract available. PMID 24232703
- [Derived] Kline JA, Hogg MM, Courtney DM, Miller CD, Jones AE, Smithline HA. D-dimer threshold increase with pretest probability unlikely for pulmonary embolism to decrease unnecessary computerized tomographic pulmonary angiography. J Thromb Haemost. 2012 Apr;10(4):572-81. doi: 10.1111/j.1538-7836.2012.04647.x. PMID 22284935
- [Derived] Kline JA, Hogg MM, Courtney DM, Miller CD, Jones AE, Smithline HA, Klekowski N, Lanier R. D-dimer and exhaled CO2/O2 to detect segmental pulmonary embolism in moderate-risk patients. Am J Respir Crit Care Med. 2010 Sep 1;182(5):669-75. doi: 10.1164/rccm.201001-0129OC. Epub 2010 May 6. PMID 20448094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I - subjects scheduled for elective surgery enrolled from January 2006-May 2006. Phase II - Hospitalized as well as Emergency Department patients were enrolled from February, 2007 to April, 2008
Groups:
- BreathScreen PE: BreathScreen PE and D-Dimer collected on subjects scheduled for elective surgery
Period: Phase II
Arm/Group | BreathScreen PE
Started | 350
Completed | 329
Not Completed | 21
Not completed — Screen Failure | 1
Not completed — Withdrawal by Subject | 1
Not completed — unable to collect blood and/or breath | 17
Not completed — Protocol Violation | 2
Period: Phase I Pre-op/Post-op
Arm/Group | BreathScreen PE
Started | 125 (The phases consisted of unique subjects. Those enrolled in Phase I did not carry over to Phase II.)
Completed | 104
Not Completed | 21

BASELINE CHARACTERISTICS:
Groups:
- Phase II: Symptomatic population undergoing testing for pulmonary embolism. Blood samples were used to obtain D-dimer levels and breath samples were used to generate the BreathScreen PE CO2/O2 ratio.
- Phase I: Pre-op/Post op subjects undergoing surgery. Blood and breath samples were collected before and after surgery. Blood samples were used to obtain D-dimer levels and breath samples were used to generate the BreathScreen PE CO2/O2 ratio.
- Total: Total of all reporting groups
Arm/Group | Phase II | Phase I | Total
Number analyzed (Participants) | 350 | 125 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (15.9) | 62 (12) | 56.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 67 | 279
  Male | 138 | 58 | 196
Region of Enrollment [Number; unit: participants]
  United States | 350 | 125 | 475

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Percentage Change in the Postoperative End Tidal CO2/O2 Ratio and D-dimer Concentration Relative to the Preoperative Measurement
Description: Median postoperative change in end tidal CO2/O2 ratio calculated as 100% * [(postoperative-preoperative)/(preoperative)]
Time Frame: Pre-op measurement: the morning of surgery. Post-op measurement: the latter of postoperative day 3 or hospital discharge
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | BreathScreen PE
Number analyzed (Participants) | 104
percent change
  end tidal CO2/O2 ratio | 0 [-13 to 16]
  D-dimer concentration | 136 [40 to 313]

2. Primary Outcome: Phase II: Probability of Pulmonary Embolism Diagnosis by D-dimer Alone vs. D-Dimer Plus CO2/O2 for Pulmonary Embolism Diagnosed by CT Scan.
Description: D-dimer > 499 ng/ml, etCO2/O2 < 0.28, Pulmonary Embolism diagnosed by CT scan
Time Frame: Measured at 45 days
Population: Completed patients minus unrecoverable data (4) and indeterminate CT scan (2).
Measure: Number; unit: probability of PE diagnosis
Groups:
- CO2/O2 Plus D-dimer: Probability of pulmonary embolism diagnosis by CO2/O2 collected with the BreathScreen PE plus D-dimer measurement as compared to D-dimer alone. D-dimer > 499 ng/ml, etCO2/O2 < 0.28, Pulmonary Embolism diagnosed by CT scan
- D-dimer: Probability of pulmonary embolism diagnosis by D-dimer alone as compared to D-dimer plus CO2/O2 measured with the BreathScren PE. D-dimer > 499 ng/ml, etCO2/O2 < 0.28, Pulmonary Embolism diagnosed by CT scan
Arm/Group | CO2/O2 Plus D-dimer | D-dimer
Number analyzed (Participants) | 323 | 323
probability of PE diagnosis | 0.32 | 0.17

ADVERSE EVENTS:
Time Frame: 45 days
Description: 348 of the 350 enrolled subjects were assessed for device-related adverse events because two participants did not have study data collection initiated: one participant requested to withdraw and another participant was designated as a screen fail.
Groups:
- Phase II: Phase II: symptomatic subjects undergoing testing for PE
- Phase I: Pre-op/Post op: subjects undergoing surgery
Arm/Group | Phase II | Phase I
Serious Adverse Events (participants affected / at risk) | 0/348 | 0/125
Other Adverse Events (participants affected / at risk) | 0/348 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No